CLINICAL TRIAL: NCT05322122
Title: Creation of Side-to-Side Compression Anastomosis Using the GT Metabolic Solutions Magnetic Anastomosis System (MAGNET System) to Achieve Duodeno-Ileostomy Diversion in Adults With Obesity and With or Without Type 2 Diabetes Mellitus
Brief Title: Creation of Side-to-Side Compression Anastomosis Using the Magnetic Anastomosis System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GT Metabolic Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTM-001
Record Dates: First submitted 2022-02-01; First posted 2022-04-11 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: An operationally seamless, 2-stage, open-label, multicenter study enrolling up to 50 subjects at up to 5 study centers across Canada and Europe:
  * Stage 1 first-in-human (FIH) and proof-of-concept with 5 subjects; and
  * Stage 2 feasibility with 45 subjects.
  There will be a pause after completing enrollment in Stage 1 to allow completion of Day 30 and evaluation of safety by the independent Data Safety Monitoring Committee (DSMB). The DSMB will confirm whether the study can advance to Stage 2. All subjects in Stage 1 and 2 will be followed for 12 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Side-to-side anastomosis duodeno-ileostomy diversion
  Interventions: Device: Side-to-side anastomosis duodeno-ileostomy diversion procedure

INTERVENTIONS:
Device: Side-to-side anastomosis duodeno-ileostomy diversion procedure — Creation of Side-to-Side Compression Anastomosis Using the GT Metabolic Solutions Magnetic Anastomosis System (The MAGNET System) to Achieve Duodeno-Ileostomy Diversion.
  Other Names: The MAGNET System

SUMMARY:
This is an operationally seamless, open-label, multicenter study enrolling up to 50 subjects with obesity and with or without type 2 diabetes at up to 5 study centers across Canada and Europe who will undergo sleeve gastrectomy (revision or de novo) with side-to-side anastomosis duodeno-ileostomy using the MAGNET System and will be followed for 12 months.

DETAILED DESCRIPTION:
The MAGNET study is an operationally seamless, 2-stage, open-label, multicenter study enrolling up to 50 subjects at up to 5 study centers across Canada and Europe as follows:

* Stage 1 first-in-human (FIH) and proof-of-concept with 5 subjects; and
* Stage 2 feasibility with 45 subjects.

There will be a pause after completing enrollment in Stage 1 to allow completion of Day 30 and evaluation of safety by the independent Data Safety Monitoring Committee (DSMB). The DSMB will confirm whether the study can advance to Stage 2. All subjects in Stage 1 and 2 will be followed for 12 months.

Study Procedure: Side-to-side anastomosis duodeno-ileostomy diversion procedure using the MAGNET System

Study Population: Adults (18 to 65 years of age, inclusive) with obesity (BMI 30-50) who meet one of the following criteria: (1) have type 2 diabetes mellitus (T2DM) or experienced weight regain following previous sleeve gastrectomy; (2) have T2DM without previous sleeve gastrectomy; or (3) are candidates for a laparoscopic single anastomosis duodenal-ileal bypass with sleeve (SADI-S) procedure and have BMI ≥ 40.

Follow-up: Each subject will return for 6 follow-up visits at Day 14, 30, 60, 90, 180, 270 and 360 (end of study).

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age, inclusive, at the time of informed consent
* BMI 30-50, inclusive with either:

  * Previous-sleeve gastrectomy (> 12 months) with either T2DM (defined as HbA1c > 6.5%) or weight regain; or
  * T2DM without previous gastrectomy; or
  * Undergoing laparoscopic single anastomosis duodenal-ileal bypass with sleeve (SADI-S) where duodeno-ileostomy is performed side to side with the MAGNET System and BMI > 40
* Agrees to refrain from any type of additional bariatric or reconstructive surgery that would affect body weight for 1 year
* If a child-bearing female, subject must commit to not becoming pregnant and agree to use contraception for 1 year
* Willing and able to comply with protocol requirements

Exclusion Criteria:

* Type 1 diabetes
* Use of injectable insulin
* Uncontrolled T2DM
* Uncontrolled hypertension, dyslipidemia or sleep apnea
* Prior intestinal, colonic or duodenal surgery, other than bariatric
* Prior surgery, trauma, prostheses, disease or genetic expression which prevent or contra- indicate the procedure, including scarring and abnormal anatomy
* Refractory gastro-esophageal reflux disease (GERD)
* Barrett's disease
* Helicobacter pylori positive and/or active ulcer disease
* Large hiatal hernia
* Inflammatory bowel or colonic diverticulitis disease
* Any anomaly precluding orogastric access by gastroscope and catheters, and manipulation techniques
* Implantable pacemaker or defibrillator
* Psychiatric disorders, except well-controlled depression with medication for >6mo, or history of substance abuse
* Woman who is either pregnant or breast feeding
* Woman of childbearing potential who does not agree to use an effective method of contraception
* Any comorbidity or current status of subject's physiological fitness that in the surgeon's or anesthesiologist's opinion represents safety concerns that make the subject medically unfit for the procedure. This includes any conditions for which endoscopic or laparoscopic surgery would be contraindicated, and any significant congenital or acquired anomalies of the GI tract at or distal to the placement of the magnets.
* Unhealed ulcers, bleeding lesions, tumor or any other lesion at target magnet deployment site
* Expected need for MR imaging within the first 2 months after the procedure
* Any anomaly preventing/contraindicating laparoscopic access and general laparoscopic procedures
* Had surgical or interventional procedure within 30 days prior to procedure
* Any scheduled surgical or interventional procedure planned within 30 days post-procedure
* Any stroke/TIA within 6 months prior to consent
* Requires chronic anticoagulation therapy (except aspirin)
* Active infections requiring antibiotic therapy, unless resolved before undergoing the study procedure
* Unable to comply with the follow-up schedule and assessments
* Recent tobacco or nicotine product cessation within < 3 months prior to informed consent
* Known allergies to the device components or contrast media
* Limited life expectancy due to terminal disease
* Currently participating in another clinical research study with an investigational drug or medical device
* A positive COVID-19 test prior to the study procedure
* Any condition that, in the investigator's opinion, may preclude completion of follow-up assessments through Day 360 (e.g., a medical condition that may increase the risk associated with study participation or may interfere with interpretation of study results, inability to adhere to the visit schedule, or poor compliance with treatment regimen)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Feasibility and performance measured by anastomosis success | Day 90
  The primary feasibility/performance endpoint is the feasibility/performance of side-to-side anastomosis duodeno-ileostomy defined as:
  * Placement of the MAGNET System (≥ 90% alignment of magnets); and
  * Passage of magnets without surgical re-intervention; and
  * Creation of a patent anastomosis, confirmed radiologically.
  The primary endpoint will be met if the feasibility/performance is confirmed in ≥ 80% of enrolled and treated subjects.

SECONDARY OUTCOMES:
To evaluate the safety of the MAGNET System | Day 30, 90, 180, and 360
  The incidence of treatment emergent AEs and SAEs is a standard measure of the safety.
  The incidence of device malfunction informs about the device reliability.
Efficacy of weight loss | Day 90, 180, and 360
  Efficacy will be assessed at Day 90, 180 and 360 based on change from baseline in total weight loss and excess weight loss (EWL)
Efficacy of metabolic improvement | Day 90, 180, and 360
  Efficacy will be assessed at Day 90, 180 and 360 based on change from baseline in functional improvement of metabolic indicators (HbA1c, blood glucose)
Quality of life improvement | Day 90, 180, and 360
  Efficacy will be assessed at Day 90, 180 and 360 based on change from baseline in quality of life improvement (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Gagner, MD, Principal Investigator — Westmount Surgical Center
Locations (4):
- CHU St Pierre, Brussels, Belgium
- Westmount Surgical Center, Westmount, Quebec, Canada
- Innova Medical Center, Tbilisi, Georgia
- Hospital Clinico San Carlos Complutense University of Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dziakova J, Torres A, Odovic M, Esteban JM, Vazquez-Romero M, Castillo A, Sanchez-Pernaute A, Gagner M. Spanish Experience with Latero-Lateral Duodeno-Ileostomy + Sleeve Gastrectomy with Magnet Anastomosis System. Obes Surg. 2024 Sep;34(9):3569-3575. doi: 10.1007/s11695-024-07432-w. Epub 2024 Aug 2. PMID 39093385
- [Derived] Gagner M, Almutlaq L, Gnanhoue G, Buchwald JN. Magnetic single-anastomosis side-to-side duodeno-ileostomy for revision of sleeve gastrectomy in adults with severe obesity: 1-year outcomes. World J Surg. 2024 Oct;48(10):2337-2348. doi: 10.1002/wjs.12304. Epub 2024 Aug 1. PMID 39090770
- [Derived] Gagner M, Abuladze D, Koiava L, Buchwald JN, Van Sante N, Krinke T. First-in-Human Side-to-Side Magnetic Compression Duodeno-ileostomy with the Magnet Anastomosis System. Obes Surg. 2023 Aug;33(8):2282-2292. doi: 10.1007/s11695-023-06708-x. Epub 2023 Jul 2. PMID 37393568